CLINICAL TRIAL: NCT06200402
Title: Antibiotic-Loaded Cement Versus Non-Antibiotic-Loaded Cement in Hip Prosthesis Surgery for Proximal Femur Fractures: A Prospective, Randomized, Single-Center, Blinded Study
Brief Title: Antibiotic-Loaded Cement Versus Non-Antibiotic-Loaded Cement in Hip Prosthesis Surgery for Proximal Femur Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Professor Giacomo Placella, Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCHIP
Record Dates: First submitted 2023-12-27; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Proximal Femoral Fractures
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): (Antibiotic-Loaded Cement Arm): This group will receive hip prosthesis surgery using antibiotic-loaded cement. The use of antibiotic-loaded cement is intended to investigate its effectiveness in reducing the rate of acute postoperative infections.
  Interventions: Drug: Antibiotic loaded
- control (Placebo Comparator): (Non-Antibiotic-Loaded Cement Arm): Participants in this group will undergo hip prosthesis surgery using non-antibiotic-loaded cement. This arm serves as the control to compare the outcomes with the antibiotic-loaded cement group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antibiotic loaded — This is the intervention for the study group. It involves the use of bone cement mixed with antibiotics (typically gentamicin or similar) in the hip prosthesis surgery. The purpose of this intervention is to assess whether the antibiotic-loaded cement reduces the incidence of postoperative infections compared to standard cement
  Arms: Intervention
Other: Placebo — Placebo
  Arms: control

SUMMARY:
The study aims to determine if antibiotic-loaded cement reduces post-surgery infection rates compared to non-antibiotic cement. The trial involves 450 elderly patients with specific hip fractures, assessing infection incidence, implant stability, and associated costs. This randomized, blinded study is conducted by IRCCS Ospedale San Raffaele.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be older than 65 years
* Fracture Type: The study includes patients with medial femoral neck fractures classified as AO type B1, B2, and B3, indicating specific types of hip fractures.
* Surgical Indication: Patients should have an indication for prosthetic hip surgery.
* Informed Consent: Patients must provide signed informed consent to participate in the study

Exclusion Criteria:

* Fracture Type: Exclusion of patients with trochanteric region fractures and femoral head fractures (AO classification types A and C), periprosthetic fractures, patients with multiple traumas or multiple fractures.
* Blood Test Anomalies: Patients with pre-operative blood test anomalies, such as ionic disorders and hemoglobin levels lower than 8 g/dL.
* Renal Insufficiency: Patients with renal insufficiency.
* Active Infections: Exclusion of patients with active infections or suspected/confirmed hypersensitivity or allergy to gentamicin, history of toxicity or reaction to aminoglycosides.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Postoperative Infections | 7 days post surgery
  This outcome measure focuses on the rate of acute infections occurring postoperatively in patients undergoing hip prosthesis surgery. The study will compare the incidence of such infections between the two groups: one receiving antibiotic-loaded cement and the other receiving non-antibiotic-loaded cement. An acute infection is typically defined based on clinical signs, laboratory markers of infection (like elevated C-reactive protein levels, white blood cell count, etc.), and the need for any additional interventions or treatments due to infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Ircss Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No